CLINICAL TRIAL: NCT07004335
Title: Efficacy and Safety of Iparomlimab and Tuvonralimab Injection in Combination With Bevacizumab After Progression on Anti-PD-(L)1 Therapy in Advanced Melanoma: A Prospective, Single-Arm, Exploratory Clinical Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhiyu Wang, MD, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025045
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: PD-(L)1; CTLA-4; Advanced Melanoma; Iparomlimab; Tuvonralimab; Bevacizumab
Keywords: Immunotherapy; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): anti PD-1/CTLA-4 (Iparomlimab/Tuvonralimab) injection and Bevacizumab
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection plus Bevacizumab

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection plus Bevacizumab — The experimental group will receive intravenous infusion of anti PD-1/CTLA-4 (Iparomlimab/Tuvonralimab) Injection (5 mg/kg) and Bevacizumab (dose 7.5mg/kg) once every 3 weeks up to 35 cycles (105 weeks).

SUMMARY:
Several studies have shown that the combination of Iparomlimab, Tuvonralimab, and Bevacizumab exhibits potent anti-tumor activity and favorable safety in various solid tumors, including liver cancer. However, the efficacy and safety of this regimen in melanoma patients with acquired resistance to immunotherapy remain unexplored and require further validation.

This study aims to evaluate the efficacy and safety of the Iparomlimab, Tuvonralimab, and Bevacizumab combination in patients with immune-resistant melanoma. Furthermore, it will analyze and compare treatment responses among different melanoma subtypes to identify optimal treatment strategies for clinical practice.

DETAILED DESCRIPTION:
This is a single-center, prospective, single-arm, exploratory clinical trial. Following the signing of informed consent, all participants will undergo screening according to the inclusion and exclusion criteria.It is anticipated that a total of 40 patients will be enrolled. Participants will receive a combination of Iparomlimab/Tuvonralimab injection and Bevacizumab every 3 weeks. Follow-up visits will be scheduled every 6 weeks. The final assessment of the study endpoints will take place at Week 105, while the last evaluation of other adverse events will be conducted at Week 109.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria for enrollment:

1. Age ≥18 years;
2. Histologically-confirmed unresectable Stage III or IV melanoma, unsuitable for local therapy;
3. Confirmed PD according to iRECIST within 12 weeks after receiving the last dose of anti-PD-(L)1 monotherapy or in combination with other treatments (including anti-CTLA-4) for at least two doses. (Up to 25% of participants may have received both anti-CTLA-4 and anti-PD-(L)1 treatment);
4. Participants with BRAF/CKIT/NRAS gene mutations must have progressed after targeted therapy;
5. Intolerant to chemotherapy or refused standard therapy;
6. Toxicity from the most recent treatment recovered to grade 1 or below (except alopecia); if participants underwent major surgery or radiotherapy >30 Gy, they must have recovered from treatment-related toxicities/complications;
7. Life expectancy of at least 3 months;
8. Eastern Cooperative Oncology Group (ECOG) score: 0-1;
9. At least one measurable lesion confirmed according to RECIST 1.1 criteria;
10. Laboratory test results at screening must meet the following requirements:

    a) Hematological tests must meet the following criteria (no blood/blood product transfusion, no correction with G-CSF or other hematopoietic stimulants within 14 days): i. Hemoglobin (Hb) ≥ 90 g/L ii. Neutrophil count (ANC) ≥ 1.5 × 10^9/L iii. Platelet count (PLT) ≥ 100×10^9/L b) Biochemical tests must meet the following criteria: i. Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN) ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 ULN (<5 ULN for participants with liver metastasis) iii. Serum creatinine (Cr) ≤ 1.5 ULN or endogenous creatinine clearance rate > 50ml/min (Cockcroft-Gault formula) iv. Urine routine test results show urine protein (UPRO) < 2+ or 24-hour urine protein quantification <1g;
11. Women of childbearing potential must have taken reliable contraceptive measures, had a negative pregnancy test (serum or urine) within 7 days before enrollment, and agree to use appropriate contraception during the trial and for 6 months after the last administration of the investigational drug. Nursing mothers should discontinue breastfeeding during the whole trial period and for 6 months after the last administration of the investigational drug to avoid the drug affecting the infant through milk. For men, they must agree to use appropriate contraception during the trial and for 120 days after the last administration of the investigational drug or have undergone surgical sterilization;
12. Provide written informed consent, and are expected to have good compliance with the study protocol.

Exclusion Criteria:

Participants meeting any of the following will be excluded:

1. Any active autoimmune disease or a history of autoimmune disease requiring treatment (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, colitis, hepatitis, pituitary炎, vasculitis, nephritis, hyperthyroidism; participants with vitiligo; childhood asthma that has completely resolved without any intervention in adulthood can be included; participants with asthma requiring bronchodilators for medical intervention cannot be included);
2. Received more than 10 mg of prednisolone or other immunosuppressive therapy within seven days prior to study treatment;
3. Severe allergic reaction to other monoclonal antibodies;
4. Uncontrolled cardiac clinical symptoms or disease, such as: heart failure of NYHA class 2 or above; unstable angina; myocardial infarction within the past year; clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; QTc >450 ms (males); QTc >470 ms (females);
5. Underwent any major surgery requiring general anesthesia within 28 days prior to the first dose;
6. Active infection, unexplained fever ≥38.5°C within seven days prior to medication, or baseline white blood cell count >15×10⁹/L; or suppurative and chronic infections, non-healing wounds;
7. With bone metastasis who received palliative radiotherapy to >5% of the bone marrow area within four weeks prior to study entry;
8. Known allergy to recombinant humanized anti-PD-(L)1 monoclonal antibody drugs, recombinant humanized anti-CTLA-4 monoclonal antibody, and/or their components;
9. Concurrent other malignancies;
10. Concurrent participation in other interventional clinical trials;
11. HIV positive; HCV positive; HBsAg or HBcAb positive with detectable HBV DNA copies (quantitative detection limit of 500 IU/ml);
12. Received live vaccine vaccination within four weeks prior to treatment initiation;
13. Ocular melanoma;
14. With active brain metastasis (previously untreated asymptomatic brain metastasis patients with ≤3 brain lesions and longest diameter <1 cm can be included. Previously treated brain metastasis patients who are clinically stable with no new or enlarged brain metastasis and have not used steroids for ≥14 days prior to study intervention can be included); other severe, acute, or chronic medical or mental disorders or laboratory abnormalities that may increase the risk associated with study participation or may interfere with the interpretation of study results, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | 105 weeks
  ORR includes complete response (CR) and partial response (PR) cases. According to RECIST V1.1, the first appearance of PR or CR requires additional imaging to confirm the lesion

SECONDARY OUTCOMES:
Overall Survival Time, OS | 105 weeks
  Overall survival (OS) is the time between the participant's first infusion injection and death from any cause.
Progression-free Survival, PFS | 105 weeks
  Progression-free survival (PFS) is defined as the time between a participant's first treatment and the first radiographic evaluation of disease progression or death from any cause, whichever comes first.
Duration of Overall Response, DOR | 105 weeks
  It was defined as the time from the first documentation of an objective response (CR or PR) to the first documentation of objective disease progression (according to RECIST v1.1 criteria) or death from any cause, whichever occurred first.

OTHER OUTCOMES:
Adverse Event, AE | 109 weeks
  The rates and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, China

IPD SHARING:
Plan to Share IPD: No